CLINICAL TRIAL: NCT04519359
Title: Novel Biomarkers Guided Stopping Nucleos(t)Ide Analogues After Long-term Virologic Suppression in CHB Patients: a Randomized Control Trial
Brief Title: Biomarkers Guided Stopping NAs Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STOP-01
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop Arm (Experimental): Stop NAs therapy
  Interventions: Other: Stop NAs therapy
- Continue Arm (No Intervention): Continue NAs therapy

INTERVENTIONS:
Other: Stop NAs therapy — Stop NAs therapy
  Arms: Stop Arm

SUMMARY:
The primary objective of this study is to evaluate hepatitis B surface antigen (HBsAg) loss in subjects who stop nucles(t)ide analogues (NAs) (Stop arm) compared to subjects who continue (Continue arm) Only subjects who already are on treatment with ETV, TDF or TAF monotherapy, and have achieved sustained virologic suppression (<20 IU/mL), HBeAg negativity, normal ALT for more than 1 year (pretreatment HBeAg + pts) or 3 years (pretreatment HBeAg - pts), plus qHBsAg <200 IU/mL, and HBV RNA or HBcrAg negativity will be included in this study. One treatment arm will stop the NAs therapy while the other treatment arm will continue the NAs therapy. Participants in the Stop arm will be monitored very closely with special focus on clinical relapse. If any participant in the Stop NAs arm exceeds one or more predefined limits for such flares or relapses, NAs treatment will be reinstituted.

ELIGIBILITY:
Key Inclusion Criteria:

* 18-65 years of old, male or female
* Chronic hepatitis B patients
* Received continuous ETV, TDF or TAF therapy for at least 1 year prior to screening and at screening
* For patients with Hepatitis B e Antigen (HBeAg)-positive at the beginning of NAs therapy, documented hepatitis B virus <20 IU/mL, HBeAg seroconversion and ALT normalization for at least 1 year prior to screening and at screening
* For patients with HBeAg-negative at the beginning of NAs therapy, documented hepatitis B virus <20 IU/mL, and ALT normalization for at least 3 year prior to screening and at screening
* <= 9 kPa on Fibroscan assessment
* qHBsAg <200 IU/mL within 24 weeks prior to screening
* HBV RNA or HBcrAg negativity within 24 weeks prior to screening

Key Exclusion Criteria:

* Experience of IFN treatment within 1 year prior to screening
* Known cirrhosis
* History of decompensated liver disease
* History of clinical hepatic decompensation in the judgement of the investigator
* Evidence of hepatocellular carcinoma
* Serological evidence of coinfection with human immunodeficiency virus (HIV), hepatitis C virus, or hepatitis D infection
* Known hypersensitivity to TDF, its metabolites, or formulation excipients
* History of malignant disease
* Lactating females
* Females wishing to became pregnant during the duration of the study
* Subjects participating in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With HBsAg Loss at Week 72 in Both Study Arms | Week 72
  HBsAg loss is defined as qualitative HBsAg result changing from positive at baseline (BL) to negative at any post-baseline visit. Proportions are based on a Kaplan-Meier estimate.

SECONDARY OUTCOMES:
Proportion of Participants With Sustained Disease Remission at Week 72 in Both Study Arms | Week 72
  Sustained Disease Remission is defined as HBeAg negativity, HBV DNA <2000 IU/mL and ALT normalization at any post-baseline visit. Proportions are based on a Kaplan-Meier estimate.
Proportion of Participants With Clinical Relapse at Week 72 in Both Study Arms | Week 72
  Clinical Relapse is defined as HBV DNA >2000 IU/mL and ALT >2 ULN at any post-baseline visit. Proportions are based on a Kaplan-Meier estimate.
Proportion of Participants With Virologic Relapse at Week 72 in Both Study Arms | Week 72
  Virologic Relapse is defined as HBV DNA >2000 IU/mL at two consecutive timepoints [at least 14 days apart] at any post-baseline visit. Proportions are based on a Kaplan-Meier estimate.
Change From Baseline in Quantitative HBsAg (IU/mL) in Both Study Arms | Week 72
  The analyses were summarized by 3 treatment subgroups: Stop NAs (NAs-Free), Restart NAs, and Continue NAs When participant randomized in the Stop NAs group restarted NAs therapy, that participant was considered part of the Restart NAs group from that point forward. For Restart NAs group, baseline is defined as the last available record on or prior to the restart date of NAs.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - No. 1 Hospital affiliated to Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fan R, Deng R, Xie Q, Wang F, Liang X, Ma H, Rao H, Gao Y, Zhong C, Guo Q, Shen S, Xu Y, Lu X, Gao H, Bai H, Dou X, Sun J. Novel HBV Biomarkers-Guided NAs Withdrawal Strategy Promotes HBsAg Clearance in Asian CHB Patients: A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2025 Sep 13:S1542-3565(25)00799-2. doi: 10.1016/j.cgh.2025.09.009. Online ahead of print. PMID 40953786